CLINICAL TRIAL: NCT04418206
Title: Validating an ELISpot for Early Detection of an Active Immune Response Against COVID-19
Acronym: EliSpot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-PP-10
Record Dates: First submitted 2020-05-18; First posted 2020-06-05 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Covid 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: COVID-19 patients will be selected in the 4 participating centres Contact subjects and healthy volunteers will be selected only in the coordinating centre (Centre Hospitalier Universitaire de Nice)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Samples With DNA (Other): Nasopharyngal swab and blood samples
  Interventions: Other: patients COVID 19

INTERVENTIONS:
Other: patients COVID 19 — Exposure to SARS-Cov2 but no symptoms (patient's family, medical staff) and General population (volunteers not exposed to SARS-Cov2)

SUMMARY:
The RT-PCR on rhino-pharynge sampling highlights the genetic material of the virus and indicates that a subject is infected with SARS-CoV-2. This test can be in about 30% of false negative cases, it does not allow to date the infection, nor to predict the asymptomatic, mild, moderate or severe evolution of the disease. In terms of public health, we need 1/ to better understand the chronology of the immune response to the virus in the general population and in contacts of index cases; 2/ To know which characteristics of the immune response are protective of future reinfections. Finally, in symptomatic subjects, we need biomarkers that predict the evolutionary mode of the disease (moderate vs. severe form).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years,
* patients with confirmed SARS-Cov2 infection (RT PCR positive)
* or patients suspected (evocative chest scanner)
* OR patients exposure to SARS-CoV2 but no symptoms (patient's family, caregivers)
* OR patients Non exposure to SARS-Cov2 volunteer subjects (general population)

Exclusion Criteria:

* pregnant or breastfeeding female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 950 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
IgA specific cells of SARS | At 7 days
  Proportion of subjects with IgA-specific cells of SARS-CoV-2's Spike 1 protein at inclusion and 7 +/-2 days later

SECONDARY OUTCOMES:
OMS progression scale | At 7 days
  The scale is 7-point ordinal.

CONTACTS AND LOCATIONS:
Overall Officials: LEROY Sylvie, Principal Investigator — CHU de Nice, pneumologie
Locations (4):
- France (4):
  - CH Antibes, Antibes, Alpes Maritimes
  - Ch Cannes, Pneumologie, Cannes, Alpes Maritimes
  - Ch Grasse, Grasse, Alpes Maritimes
  - CHU de nice, Nice, Alpes-Maritimes

IPD SHARING:
Plan to Share IPD: Undecided